CLINICAL TRIAL: NCT03830489
Title: Intensive High-volume Bowel Cleansing Regimen Versus Low-volume Bowel Regimen in Patients With a High Risk of Poor Colonic Cleansing Following a Validated Predictive Score
Brief Title: Impact of a Predictive Score of Bowel Preparation Quality in Clinical Practice
Acronym: REPREP2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Score-guided colon cleansing
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Cleansing Quality of the Colon
Keywords: Cleansing quality score; Colonoscopy
MeSH Terms: interventions — Polyethylene Glycols; Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Only the endoscopists in charge of rating the bowel cleansing during the colonoscopy will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Large volume based preparation (Experimental): This strategy will consist of split dose 4 L polyethylene glycol plus 10 mg bisacodyl plus 3 days of fiber-free diet.
  Interventions: Drug: polyethylene glycol
- Low volume based preparation (Active Comparator): This strategy will consist of split dose 2 L polyethylene glycol plus Ascorbic acid plus 1 day of fiber-free diet
  Interventions: Drug: polyethylene glycol plus ascorbic acid

INTERVENTIONS:
Drug: polyethylene glycol — The experimental arm will take 4 L polyethylene glycol solution (PEG) in split dose plus bisacodyl and 3 days of fiber-free diet
  Arms: Large volume based preparation
Drug: polyethylene glycol plus ascorbic acid — The control arm will take 2 L polyethylene glycol solution (PEG) plus ascorbic acid in split dose plus 1 day of fiber-free diet
  Arms: Low volume based preparation

SUMMARY:
This is a single center randomized controlled trial to compare the colon cleansing quality determined by the Boston Bowel Preparation Scale achieved by two strategies in patients with high risk of poor colon cleansing defined as those patients with a score> 1.225 following a predictive score previously published: one group will receive an intensified split-dose 4 L polyethylene glycol solution (PEG) plus bisacodyl and 3 days of fiber-free diet and the other group a split-dose 2 L PEG solution with ascorbic plus bisacodyl and 1 day of fiber-free diet.

Patients with a score ≤ 1.225 will receive a split-dose 2 L PEG solution with ascorbic plus bisacodyl and 1 day of fiber-free diet.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blind phase IV study in which all outpatients scheduled for a colonoscopy will be given a different bowel cleansing strategy (conventional or intensified) according to a scoring system already validated in the investigator's center, designed with variables independently associated with poor bowel cleansing, constipation, abdominal/pelvic surgery, comorbidity and to be on antidepressant treatment. According to this system, a score equal to or less than 1.225, predicts with a high confidence (negative predictive value = 88%) a suitable cleansing quality with a standard preparation protocol. Therefore, these subjects will be advised of a conventional preparation (low fiber diet the day before the examination and low volume preparation consisting of 2 L of PEG with ascorbic acid). Subjects with a score greater than 1.225 will be randomized to receive an intensive bowel preparation (low fiber diet three days prior to colonoscopy and large bowel preparation consisting of 4 L PEG with bisacodyl) or a conventional one (low fiber diet the day before the examination and 2 L of PEG with ascorbic acid). The choice of low-volume preparation as a control is supported by the absence of significant differences in quality of cleanliness in patients with a score > 1.225 among patients prepared with high or low volume and that low volume preparation appears to improve tolerance and compliance.

A researcher will offer to participate in the study to all outpatients with a scheduled colonoscopy, who meet all the inclusion criteria and none of the exclusion criteria. The researchers will explain the purpose of the study and will ask to sign the informed consent. They will give verbal and written information on the bowel preparation strategy. Thus, according to the allocation group, participants must comply with a large volume cleansing strategy or a conventional one. For patients with a low score (≤ 1.225) a conventional preparation will be recommended.

Patients must complete a baseline questionnaire at the inclusion visit and another questionnaire at the colonoscopy visit.

The hypothesis of the study is that in patients with a high risk of poor bowel preparation, the large bowel based preparation strategy is superior to the conventional bowel preparation in achieving an acceptable bowel cleansing assessed by a validated scale (Boston Bowel Preparation Score).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Outpatient colonoscopy
* Willing to participate (informed consent signed).

Exclusion Criteria:

* Intestinal perforation
* Poorly controlled arterial hypertension (HTAS> 180 HTAD> 100)
* Congestive heart failure
* NYHA III-IV
* Acute hepatic failure
* End-stage renal disease (creatinine <15 ml / min dialysis or pre-dialysis)
* Pregnancy or breastfeeding
* Known hypersensitivity reaction to drug components
* Phenylketonuria or Glucose-6-phosphate dehydrogenase deficiency
* Dementia with difficulty in intake of Preparation
* Past history of poor bowel preparation colonic cleanliness
* Inability to follow the instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale | 8 months
  This scale goes from 0 (no preparation) to 3 points (excellent preparation) in the three segments of the colon (proximal, transverse and distal). The maximum score is 9 points

SECONDARY OUTCOMES:
Proportion of polyps detected in each arm | 8 months
  Number of polyps in one arm/total of polyps detected
Tolerance to bowel preparation | 8 months
  It will be subjective and assessed by a visual analog scale (0 very bad, 10 excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Goretti Hernandez, MD, Principal Investigator — Hospital Universitario de Canarias
Locations (1):
- Department of Gastroenterology, San Cristóbal de La Laguna, S/C de Tenerife, Spain

REFERENCES:
- [Result] Gimeno-Garcia AZ, Hernandez G, Aldea A, Nicolas-Perez D, Jimenez A, Carrillo M, Felipe V, Alarcon-Fernandez O, Hernandez-Guerra M, Romero R, Alonso I, Gonzalez Y, Adrian Z, Moreno M, Ramos L, Quintero E. Comparison of Two Intensive Bowel Cleansing Regimens in Patients With Previous Poor Bowel Preparation: A Randomized Controlled Study. Am J Gastroenterol. 2017 Jun;112(6):951-958. doi: 10.1038/ajg.2017.53. Epub 2017 Mar 14. PMID 28291237
- [Result] Gimeno-Garcia AZ, Baute JL, Hernandez G, Morales D, Gonzalez-Perez CD, Nicolas-Perez D, Alarcon-Fernandez O, Jimenez A, Hernandez-Guerra M, Romero R, Alonso I, Gonzalez Y, Adrian Z, Carrillo M, Ramos L, Quintero E. Risk factors for inadequate bowel preparation: a validated predictive score. Endoscopy. 2017 Jun;49(6):536-543. doi: 10.1055/s-0043-101683. Epub 2017 Mar 10. PMID 28282690
- [Result] Dik VK, Moons LM, Huyuk M, van der Schaar P, de Vos Tot Nederveen Cappel WH, Ter Borg PC, Meijssen MA, Ouwendijk RJ, Le Fevre DM, Stouten M, van der Galien O, Hiemstra TJ, Monkelbaan JF, van Oijen MG, Siersema PD; Colonoscopy Quality Initiative. Predicting inadequate bowel preparation for colonoscopy in participants receiving split-dose bowel preparation: development and validation of a prediction score. Gastrointest Endosc. 2015 Mar;81(3):665-72. doi: 10.1016/j.gie.2014.09.066. Epub 2015 Jan 17. PMID 25600879
- [Result] Hassan C, Fuccio L, Bruno M, Pagano N, Spada C, Carrara S, Giordanino C, Rondonotti E, Curcio G, Dulbecco P, Fabbri C, Della Casa D, Maiero S, Simone A, Iacopini F, Feliciangeli G, Manes G, Rinaldi A, Zullo A, Rogai F, Repici A. A predictive model identifies patients most likely to have inadequate bowel preparation for colonoscopy. Clin Gastroenterol Hepatol. 2012 May;10(5):501-6. doi: 10.1016/j.cgh.2011.12.037. Epub 2012 Jan 10. PMID 22239959
- [Derived] Gimeno-Garcia AZ, Benitez-Zafra F, Hernandez A, Hernandez-Negrin D, Nicolas-Perez D, Hernandez G, Baute-Dorta JL, Cedres Y, Del-Castillo R, Mon J, Jimenez A, Navarro-Davila MA, Rodriguez-Hernandez E, Alarcon O, Romero R, Felipe V, Segura N, Hernandez-Guerra M. Agreement between the perception of colon cleansing reported by patients and colon cleansing assessed by a validated colon cleansing scale. Gastroenterol Hepatol. 2024 Feb;47(2):130-139. doi: 10.1016/j.gastrohep.2023.02.009. Epub 2023 Mar 2. English, Spanish. PMID 36870478
- [Derived] Gimeno-Garcia AZ, Hernandez G, Baute Dorta JL, Reygosa C, de la Barreda R, Hernandez-Bustabad A, Amaral C, Cedres Y, Del Castillo R, Nicolas-Perez D, Jimenez A, Alarcon-Fernandez O, Hernandez-Guerra M, Romero R, Alonso I, Gonzalez Y, Adrian Z, Hernandez D, Ramos L, Carrillo M, Felipe V, Hernandez A, Rodriguez-Jimenez C, Quintero E. An Enhanced High-Volume Preparation for Colonoscopy Is Not Better Than a Conventional Low-Volume One in Patients at Risk of Poor Bowel Cleansing: A Randomized Controlled Trial. Front Med (Lausanne). 2021 Mar 22;8:654847. doi: 10.3389/fmed.2021.654847. eCollection 2021. PMID 33829030